CLINICAL TRIAL: NCT02224001
Title: A New Concept in the Tip Plasty of Asian Rhinoplasty : The Flag Technique by Use of Only A Septal Cartilage Without Septal Extension Grafts
Brief Title: A New Concept in the Tip Plasty of Asian Rhinoplasty
Acronym: TP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winners Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tip Plasty
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Asian Rhinoplasty
Keywords: tip plasty; septal cartilage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asian rhinoplasty, septal cartilage (Experimental): A New Concept in the Tip Plasty of Asian Rhinoplasty : The Flag Technique by Use of Only A Septal Cartilage without Septal Extension Grafts
  The investigators propose the new technique, so called 'Flag Technique' by a tip-strut complex in a flag-like shape : using only the septal cartilage as an elongated columellar septal strut graft, a shield graft , bilateral mini-spreader grafts of the upper part in the elongated columellar septal strut graft without the septal extension graft to achieve the desired the result.
  Interventions: Procedure: The Flag Technique

INTERVENTIONS:
Procedure: The Flag Technique — A New Concept in the Tip Plasty of Asian Rhinoplasty : The Flag Technique by Use of Only A Septal Cartilage without Septal Extension Grafts
  The investigators propose the new technique, so called 'Flag Technique' by a tip-strut complex in a flag-like shape : using only the septal cartilage as an elongated columellar septal strut graft, a shield graft , bilateral mini-spreader grafts of the upper part in the elongated columellar septal strut graft without the septal extension graft to achieve the desired the result.

SUMMARY:
For achieving the desired refinements in Asian patients, sufficient septal cartilage must be needed for the ieal tip projection and lengthening of the nose by the septal extension graft, columellar septal strut graft, and onlay tip graft, shield graft. Actually there are many cases having insufficient septal cartilages in Asian augmentation rhinoplasty.

The investigators propose the new technique, so called 'Flag Technique' by a tip-strut complex in a flag-like shape : using only the septal cartilage as an elongated columellar septal strut graft, a shield graft , bilateral mini-spreader grafts of the upper part in the elongated columellar septal strut graft without the septal extension graft to achieve the desired the result.

DETAILED DESCRIPTION:
The investigators propose the new technique, so called 'Flag Technique' by a tip-strut complex in a flag-like shape : using only the septal cartilage as an elongated columellar septal strut graft, a shield graft , bilateral mini-spreader grafts of the upper part in the elongated columellar septal strut graft without the septal extension graft to achieve the desired the result.

ELIGIBILITY:
Inclusion Criteria:

* primary case
* secondary case

Exclusion Criteria:

* septal cartilage harvested state
* congenital anomaly in septal cartilage

Ages: 17 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | six months
  * tip deviation : 1 case
  * low tip projection : 1 case

CONTACTS AND LOCATIONS:
Overall Officials: CHEOLHWAN KIM, MD, Principal Investigator — Winners Clinic
Locations (1):
- The Department of Plastic Surgery, Winners Clinic, Gangnamgu, Seoul, South Korea

REFERENCES:
- [Background] 1.Toriumi, D.M. Augmentation rhinoplasty with autologous cartilage grafting. In Park JI, Toriumi, D.M., eds. Asian Facial Cosmetic Surgery. Philadelphia: Saunders-Elsvier, 2007. 2.Toriumi, D.M. Autologous grafts are worth the extra time. Arch Otolaryngol Head Neck Surg 126:562-564, 2000. 3.Toriumi, D.M., DeRosa J. The Asian nose. In R. J. Rohrich, W. P. Jr. Adams, and J. Ahmad, J. P. Gunter (Eds.), Dallas Rhinoplasty: Nasal Surgery by the Masters, Vol 2, 3rd Ed. St. Louise: Quality Medical, 2014. Pp. 1226-1229. 4.Byrd , H.S., Burt, J.D., Andochick, S., et al. Septal extension grafts: a method for controlling tip projection and shape. Plast Reconstr Surg 100:999-1010, 1997. 5.Rohrich R.J., Kurkjian T.J., Hoxworth R.E., et al. The effect of the columellar strut graft on the nasal tip position in primary rhinoplasty. Plast Reconstr Surg 130:926-932, 2012. Erratum in Plast Reconstr Surg 130:1399, 2012.